CLINICAL TRIAL: NCT06246617
Title: A Real-World Study to Evaluate the Clinical Performance and Safety of da Vinci SP Surgical System for Single-Port Thoracic Surgeries
Brief Title: Valuate the Clinical Performance and Safety of da Vinci SP Surgical System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-020
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-11

CONDITIONS: da Vinci SP Surgical System; Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: Subjects who have received or plan to receive pulmonary lobectomy/segmentectomy, mediastinal tumor resection (including thymectomy), radical resection of esophagus cancer or other surgeries with the SP single-port robot
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Arm 1 (Experimental): Subjects who have received or plan to receive pulmonary lobectomy/segmentectomy, mediastinal tumor resection (including thymectomy), radical resection of esophagus cancer or other surgeries with the SP single-port robot.
  Interventions: Device: da Vinci SP Surgical System for Single-Port Thoracic Surgeries

INTERVENTIONS:
Device: da Vinci SP Surgical System for Single-Port Thoracic Surgeries — Subjects who have received or plan to receive pulmonary lobectomy/segmentectomy, mediastinal tumor resection (including thymectomy), radical resection of esophagus cancer or other surgeries with the SP single-port robot.

SUMMARY:
This clinical trial is a real-world study to evaluate the clinical performance and safety of da Vinci SP Surgical System ("SP single-port robot" for short) for single-port robot-assisted thoracic surgeries in the real world, providing a real world evidence for clinical application of the product in the Chinese population.

DETAILED DESCRIPTION:
Subjects who have received or plan to receive pulmonary lobectomy/segmentectomy, mediastinal tumor resection (including thymectomy), radical resection of esophagus cancer or other surgeries with the SP single-port robot.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who have received or plan to receive pulmonary lobectomy/segmentectomy, mediastinal tumor resection (including thymectomy), radical resection of esophagus cancer or other surgeries with the SP single-port robot; 2. Patients who voluntarily decide to participate in the study and sign the ICF (or exempt from signature of the ICF as approved by the EC).

Exclusion Criteria:

* 1. Patients with missing data on the primary endpoint in retrospective cases; 2. Subjects having any contraindications of single-port robot surgery; 3. The intraoperative anatomy determined that minimally invasive surgery was not suitable; 4. Patients who are considered inappropriate to participate in this study by investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
Intraoperative conversion rate | intraoperative
  Intraoperative conversion rate = number of subjects with intraoperative conversion/total number of subjects ×100%.
  The intraoperative conversion is defined as conversion to other procedures (including but not limited to traditional laparoscopic surgeries, other robot-assisted surgeries, open surgeries and so on) for various reasons during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Li C, Chen X, Wang X, Guo W, Zhang Y, Chen F, Li H. Single-Port Robotic-Assisted Approach in Thoracic Surgery: A Prospective Real-World Study. Interdiscip Cardiovasc Thorac Surg. 2025 Jul 3;40(7):ivaf161. doi: 10.1093/icvts/ivaf161. PMID 40658465